CLINICAL TRIAL: NCT01502410
Title: A Phase II Study of the Raf Kinase and Receptor Tyrosine Kinase Inhibitor Sorafenib in Children and Young Adults With Relapsed/Refractory Rhabdomyosarcoma, Wilms Tumor, Hepatocellular Carcinoma, and Papillary Thyroid Carcinoma
Brief Title: Sorafenib Tosylate in Treating Younger Patients With Relapsed or Refractory Rhabdomyosarcoma, Wilms Tumor, Liver Cancer, or Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00106; NCI-2012-00106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL1121 (Other: Children's Oncology Group); CDR0000721611 (Other: ClinicalTrials.gov); ADVL1121 (Other: Children's Oncology Group); ADVL1121 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Childhood Hepatocellular Carcinoma; Papillary Thyroid Cancer; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Childhood Liver Cancer; Recurrent Childhood Rhabdomyosarcoma; Recurrent Thyroid Cancer; Recurrent Wilms Tumor and Other Childhood Kidney Tumors
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid Neoplasms; Wilms Tumor | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 Relapsed/Refractory Rhabdomyosarcoma (Experimental): Patients with relapsed or refractory rhabdomyosarcoma receive sorafenib tosylate PO BID on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  sorafenib tosylate: Given PO dosage 200 mg/m2/dose (max dose:400 mg/dose) given every 12 hours on days 1-28
  pharmacological study: Optional correlative studies
  laboratory biomarker analysis: Optional correlative studies
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study; Other: laboratory biomarker analysis
- Group 2 Relapsed/Refractory Wilms tumor (Experimental): Patients with relapsed or refractory Wilms tumor receive sorafenib tosylate PO BID on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  sorafenib tosylate: Given PO dosage 200 mg/m2/dose (max dose:400 mg/dose) given every 12 hours on days 1-28
  pharmacological study: Optional correlative studies
  laboratory biomarker analysis: Optional correlative studies
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study; Other: laboratory biomarker analysis
- Group 3 Relapsed/Refractory hepatocellular carcinoma (Experimental): Patients with relapsed or refractory hepatocellular carcinoma receive sorafenib tosylate PO BID on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  sorafenib tosylate: Given PO dosage 200 mg/m2/dose (max dose:400 mg/dose) given every 12 hours on days 1-28
  pharmacological study: Optional correlative studies
  laboratory biomarker analysis: Optional correlative studies
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study; Other: laboratory biomarker analysis
- Group 4 Papillary thyroid carcinoma (Experimental): Patients with relapsed or refractory papillary thyroid carcinoma receive sorafenib tosylate PO BID on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  sorafenib tosylate: Given PO dosage 200 mg/m2/dose (max dose:400 mg/dose) given every 12 hours on days 1-28
  pharmacological study: Optional correlative studies
  laboratory biomarker analysis: Optional correlative studies
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO dosage 200 mg/m2/dose (max dose:400 mg/dose) given every 12 hours on days 1-28
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: pharmacological study — Optional correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II trial studies how well sorafenib tosylate works in treating younger patients with relapsed or refractory rhabdomyosarcoma, Wilms tumor, liver cancer, or thyroid cancer. Sorafenib tosylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate to sorafenib tosylate (sorafenib) in children with relapsed or refractory rhabdomyosarcoma, Wilms tumor, hepatocellular carcinoma (HCC), or papillary thyroid carcinoma (PTC).

SECONDARY OBJECTIVES:

I. To further define and describe the toxicities of sorafenib administered on an oral, twice-daily continuous schedule.

II. To further characterize the pharmacokinetics of sorafenib in children with refractory cancer.

III. To estimate the progression-free survival on sorafenib for rhabdomyosarcoma, Wilms tumor, and hepatocellular carcinoma and compare to a group of patients enrolled on selected closed Phase II studies of Children Oncology Group (COG).

IV. To assess the biologic activity of sorafenib on vascular endothelial growth factor (VEGF) and soluble vascular endothelial growth factor receptor-2 (VEGFR-2) in peripheral blood samples. (Exploratory) V. To evaluate the presence of BRAF mutations and RET/PTC rearrangements in patients with PTC. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to diagnosis (rhabdomyosarcoma vs Wilms tumor vs hepatocellular carcinoma vs papillary thyroid carcinoma).

Patients receive sorafenib tosylate orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and periodically during study for pharmacokinetic studies, and VEGF and VEGFR-2 analysis by ELISA. Previously collected formalin-fixed paraffin-embedded tissue samples, from patients with papillary thyroid carcinoma, are also analyzed for BRAF mutation and RET/PTC rearrangements by PCR.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of one of the malignancies listed below at original diagnosis or at relapse:

  * Rhabdomyosarcoma (RMS)
  * Wilms tumor
  * Hepatocellular carcinoma (HCC)
  * Papillary thyroid carcinoma (PTC)
* Patients must have relapsed or refractory disease (RMS, Wilms tumor, HCC, PTC)

  * Patients must have radiographically measurable disease; measurable disease is defined as the presence of at least one lesion on magnetic resonance imaging (MRI) or computed tomography (CT) scan that can be accurately measured with the longest diameter a minimum of 10 mm in at least one dimension (CT scan slice thickness no greater than 5 mm)

    * The following do not qualify as measurable disease:

      * Malignant fluid collections (e.g., ascites, pleural effusions)
      * Bone marrow infiltration
      * Lesions only detected by nuclear medicine studies (e.g., bone, gallium, or positron emission tomography [PET] scans)
      * Elevated tumor markers in plasma or cerebrospinal fluid(CSF)
      * Previously radiated lesions that have not demonstrated clear progression post radiation
      * Leptomeningeal lesions that do not meet the requirements noted above
* Patients with HCC must be relapsed or refractory to conventional chemotherapy
* Patients with PTC must be refractory to radioactive iodine (RAI)
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Patients with known metastasis to the brain will be excluded from trial participation unless treated surgically or with radiotherapy and stable with no recurrent lesions for at least 3 months
* Rhabdomyosarcoma and Wilms strata: patients must be ≥ 24 months and ≤ 30 years of age at study enrollment
* Hepatocellular carcinoma (HCC): patients must be ≥ 24 months and < 18 years of age at study enrollment
* Papillary thyroid carcinoma (PTC): patients must be ≥ 24 months and ≤ 21 years of age at study enrollment
* Patients must have a Lansky or Karnofsky performance status score of ≥ 50%, corresponding to ECOG categories 0, 1, or 2

  * Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age
  * Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Peripheral absolute neutrophil count (ANC) ≥ 1,000/μL
* Platelet count ≥ 75,000/μL (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment)
* Hemoglobin 8.0 g/dL (may receive red blood cell[RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate(GFR) 70 mL/min OR a serum creatinine based on age/gender as follows:

  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (≥ 16 years of age)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* SGPT (ALT) ≤ 135 U/L (for the purpose of this study, the ULN for SGPT is 45 U/L)
* PT, PTT, and INR < 1.5 times ULN
* Normal serum lipase and amylase (per institutional normal values)
* No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination
* A blood pressure (BP) ≤ the 95^th percentile for age, height, and gender; and not receiving medication for treatment of hypertension
* Patients who are pregnant or breast-feeding are not eligible
* Negative pregnancy tests must be obtained in girls who are post-menarchal
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method beginning at the signing of the informed consent until at least 30 days after the last dose of the study drug
* Patients with clinical symptoms of hepatic encephalopathy or ascites are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients with evidence of bleeding diathesis are not eligible
* Patients with known Gilbert syndrome are not eligible
* Patients who, in the opinion of the investigator, may not be able to comply with the safety-monitoring requirements of the study are not eligible
* No concurrent chemotherapy, radiation therapy, immunomodulating agents, or other investigational agents
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Patients with solid tumors must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
* At least 7 days must have elapsed since the completion of therapy with a growth factor (at least 14 days must have elapsed after receiving pegfilgrastim)
* At least 7 days must have elapsed since completion of therapy with a biologic agent;

  * For agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur
* At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody
* At least 2 weeks must have elapsed since local palliative radiotherapy (XRT) (small port); ≥ 3 months must have elapsed if prior craniospinal XRT was received, if ≥ 50% of the pelvis was irradiated, or if TBI was received; ≥ 6 weeks must have elapsed if other substantial bone marrow irradiation was given
* No evidence of active graft-vs-host disease and ≥ 2 months must have elapsed since transplant (stem cell transplant or rescue without total-body irradiation)
* For patients with papillary thyroid carcinoma (PTC) only: ≥ 3 weeks from prior radioiodine (RAI) treatment
* Patients requiring corticosteroids that have not been on a stable or decreasing dose of corticosteroid for 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post transplant are not eligible for this trial
* Patients who take cytochrome P450 enzyme-inducing anti-epileptic drugs (phenytoin, carbamazepine, or phenobarbital), rifampin, grapefruit juice, or St. Johns wort will not be eligible for the trial
* Patients who have received prior treatment with sorafenib are not eligible
* Patients must not be on therapeutic anti-coagulation;

  * Prophylactic anticoagulation (i.e., low-dose warfarin) of venous or arterial devices is allowed provided that the requirements for prothrombin time(PT), partial thromboplastin time(PTT), and international normalized ratio(INR) are met

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, MD, Principal Investigator — Children's Oncology Group
Locations (92):
- United States (83):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Childrens Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Mark O Hatfield-Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (7):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only Rhabdomyosarcoma and Wilms Tumor patients are reported as there were no accruals on Hepatocellular carcinoma and no accruals on Thyroid carcinoma.
Period: Overall Study
Arm/Group | Group 1 Relapsed/Refractory Rhabdomyosarcoma | Group 2 Relapsed/Refractory Wilms Tumor | Group 3 Relapsed/Refractory Hepatocellular Carcinoma | Group 4 Papillary Thyroid Carcinoma
Started | 10 | 10 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 10 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Lack of Efficacy | 7 | 7 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Relapsed/Refractory Rhabdomyosarcoma | Group 2 Relapsed/Refractory Wilms Tumor | Group 3 Relapsed/Refractory Hepatocellular Carcinoma | Group 4 Papillary Thyroid Carcinoma | Total
Number analyzed (Participants) | 10 | 10 | 0 | 0 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 10 |  |  | 17
  Between 18 and 65 years | 3 | 0 |  |  | 3
  >=65 years | 0 | 0 |  |  | 0
Age, Continuous [Median (Full Range); unit: years] | 12 [5 to 21] | 10.5 [7 to 18] |  |  | 11 [5 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 |  |  | 9
  Male | 6 | 5 |  |  | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 |  |  | 2
  Not Hispanic or Latino | 10 | 8 |  |  | 18
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 0 | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 3 | 0 |  |  | 3
  White | 7 | 7 |  |  | 14
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 2 |  |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 |  |  | 19
  Canada | 1 | 0 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response by RECIST Criteria v 1.1
Description: Response rates will be calculated as the number of evaluable patients who are responders. Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR): Disappearance of all target lesions, Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD, Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started and Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 6 cycles (168 days)
Population: Only Rhabdomyosarcoma and Wilms Tumor patients are included in this analysis as there were no accruals on Hepatocellular carcinoma and no accruals on Thyroid carcinoma.
Measure: Number; unit: participants
Arm/Group | Group 1 Relapsed/Refractory Rhabdomyosarcoma | Group 2 Relapsed/Refractory Wilms Tumor
Number analyzed (Participants) | 10 | 10
participants
  Non-Responder | 10 | 10
  Responder | 0 | 0

2. Secondary Outcome: Progression-free Survival According to RECIST Version 1.1
Description: Percent probability of being progression free six months following enrollment. Progression-free interval (PFI) will be calculated as the date of enrollment until the end PFI date, where that date is calculated as the date of disease progression, date of death, date of removal of all tumors by surgery or last patient contact, whichever occurs first.
Time Frame: Six months after enrollment
Population: All eligible patients are included in this analysis for both Rhabdomyosarcoma and Wilms Tumor. However, there were no accruals on the disease arms for Hepatocellular carcinoma and Papillary Thyroid carcinoma and were not included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Group 1 Relapsed/Refractory Rhabdomyosarcoma | Group 2 Relapsed/Refractory Wilms Tumor
Number analyzed (Participants) | 10 | 10
percentage of probability | 10 [0.57 to 36] | 23 [3.5 to 52]

3. Secondary Outcome: The Number of Patients Who Experience at Least One Grade 3 or Higher CTC Version 4 Toxicity,
Description: Each patient is classified as having experienced grade 3 or higher CTC version 4 toxicity if at any time during protocol therapy such an event is observed for the individual.
Time Frame: six cycles of chemotherapy; expected to be 126 days of treatment
Population: All eligible patients diagnosed with Rhabdomyosarcoma or Wilms Tumor are combined in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Rhabdomyosarcoma and Wilms Tumor: These are the responses of the patient's organs to the drug. As such, these measures are unrelated to the particular diagnosed disease. Therefore, both Rhabdomyosarcoma and Wilms Tumor are combined in this analysis.
Arm/Group | Rhabdomyosarcoma and Wilms Tumor
Number analyzed (Participants) | 20
Participants | 14

4. Secondary Outcome: Pharmacokinetic (PK) Parameters of Sorafenib Tosylate
Description: The trough sorafenib concentration is evaluated at baseline (prior to administration of Sorafenib) and 12 hours after administration of Sorafenib on day 15, day 56, day 112 and day 168 in micrograms/ml.
Time Frame: Prior to administration of Sorafenib (baseline), day 15, day 56, day 112 and day 168
Population: Baseline sample was available for only 9 participants.
Measure: Mean (Full Range); unit: micrograms/ml
Groups:
- Rhabdomyosarcoma and Wilms Tumor: Serum concentration are the responses of the patient's organs to the drug. As such, these measures are unrelated to the particular disease with which the patient was diagnosed and were combined for analysis.
Arm/Group | Rhabdomyosarcoma and Wilms Tumor
Number analyzed (Participants) | 9
micrograms/ml
  Baseline | 0 [0 to 0]
  Day 15 of protocol therapy | 6.51 [0.09 to 13.64]
  Day 56 of protocol therapy: number analyzed (Participants) | 4
  Day 56 of protocol therapy | 6.99 [3.33 to 10.10]
  Day 112 of protocol therapy: number analyzed (Participants) | 1
  Day 112 of protocol therapy | 4.10 [4.10 to 4.10]
  Day 168 of protocol therapy: number analyzed (Participants) | 1
  Day 168 of protocol therapy | 5.20 [5.20 to 5.20]

5. Secondary Outcome: Change in VEGF and VEGFR-2
Description: Serum VEGF and VEGF receptor 2 Concentration is evaluated at baseline and at day 15 of protocol therapy in picograms/ml.
Time Frame: Prior to the administration of sorafenib (baseline) and day 15 of protocol therapy
Population: Change in VEGF and VEGFR-2 are the responses of the patient's organs to the drug. As such, these measures are unrelated to the particular disease with which the patient was diagnosed, and were combined for analysis.
Measure: Mean (Full Range); unit: picograms/ml
Arm/Group | Rhabdomyosarcoma and Wilms Tumor
Number analyzed (Participants) | 9
picograms/ml
  VEGF Baseline | 155.75 [28.01 to 452.22]
  VEGF Day 15 | 209.92 [70.10 to 470.38]
  VEGF-R2 Baseline | 9594.04 [651.8 to 15576.39]
  VEG-R2 Day 15 | 7948.48 [5569.73 to 11637.18]

6. Secondary Outcome: Presence of BRAF Mutation or RET/PTC Rearrangement
Description: Descriptive statistics including mean, median, standard deviation, and range will be calculated for baseline for patients with PTC, TG and TG antibody, and presence of BRAF mutation or RET/PTC rearrangement.
Time Frame: At baseline
Population: No patients were enrolled with PTC (papillary thyroid carcinoma) so there are no patients who can contribute to this outcome measure.
Arm/Group | Group 1 Relapsed/Refractory Rhabdomyosarcoma | Group 2 Relapsed/Refractory Wilms Tumor
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: SAE field contains NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Only Grade 3 and higher Adverse Events were collected/assessed in this study.
Groups:
- Group 1 Relapsed/Refractory Rhabdomyosarcoma: Patients with relapsed or refractory rhabdomyosarcoma receive sorafenib tosylate PO BID on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
- Group 2 Relapsed/Refractory Wilms Tumor: Patients with relapsed or refractory Wilms tumor receive sorafenib tosylate PO BID on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Group 1 Relapsed/Refractory Rhabdomyosarcoma | Group 2 Relapsed/Refractory Wilms Tumor
Serious Adverse Events (participants affected / at risk) | 4/10 | 3/10
Other Adverse Events (participants affected / at risk) | 5/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Relapsed/Refractory Rhabdomyosarcoma (N=10) | Group 2 Relapsed/Refractory Wilms Tumor (N=10)
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pain (General disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Relapsed/Refractory Rhabdomyosarcoma (N=10) | Group 2 Relapsed/Refractory Wilms Tumor (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less